CLINICAL TRIAL: NCT05295420
Title: The Role of Platelet Rich Plasma Injections in Cases of Stress Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Collaborators: Al-Azhar University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ahmed Tahoon
Record Dates: First submitted 2022-02-27; First posted 2022-03-25 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Stress Urinary Incontinence; Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- platelet-rich plasma (Experimental): to assess the role of platelet-rich plasma in the treatment of SUI as a non-invasive method
  Interventions: Procedure: platelet rich plasma

INTERVENTIONS:
Procedure: platelet rich plasma — Injection of Platelet Rich Plasma in the female conditions that suffer from SUI

SUMMARY:
Urinary incontinence can impact on one's social, physical, mental, and sexual wellbeing, and lead to depression and social isolation Stress urinary incontinence (SUI) refers to the involuntary leakage of urine accompanying physical exertion (i.e. coughing, exercise, and sneezing). It is commonly acquired after pregnancy and childbirth due to the weakening of the pelvic floor muscles that support the urethra against the anterior vaginal wall.

Current SUI treatment includes surgery to re-establish sufficient urethral resistance in order to prevent urine leakage during increased intra-abdominal pressure.

DETAILED DESCRIPTION:
Urinary incontinence can impact on one's social, physical, mental, and sexual wellbeing, and lead to depression and social isolation.

Stress urinary incontinence (SUI) refers to the involuntary leakage of urine accompanying physical exertion (i.e. coughing, exercise, and sneezing). It is commonly acquired after pregnancy and childbirth due to the weakening of the pelvic floor muscles that support the urethra against the anterior vaginal wall.

Current SUI treatment includes surgery to re-establish sufficient urethral resistance in order to prevent urine leakage during increased intra-abdominal pressure.

The mid-urethral sling (MUS) has become the preferred procedure, as it is less invasive than the Burch colposuspension. However, the MUS procedure has a 5-20% failure rate and carries risks such as infection, voiding dysfunction, hemorrhage, pain, bladder or urethral injury, and mesh erosion.

Hence, there is a need for alternative efficacious, outpatient SUI treatments. Platelet-derived therapies are a growing trend across multiple medical and surgical specialties. Evidence suggests that platelets play an important role in tissue repair, vascular remodeling and inflammatory and immune responses through secretion of growth factors, cytokines, and chemokines.

These biologically active proteins include transforming growth factor-β, platelet-derived growth factor, platelet-derived epithelial growth factor, insulin-like growth factor, vascular endothelial growth factor. These growth factors are implicated in many aspects of natural wound healing, including chemotaxis, cell proliferation, cell differentiation. The key role of platelets in these processes makes them an attractive candidate for therapies aimed at accelerating natural healing.

One of the most well-described platelet-based therapies is autologous platelet-rich plasma (PRP). PRP is derived from the centrifugation of whole blood with a separator gel to remove the red and white blood cells. The resulting supernatant has a greater than four-fold increase in platelets and other plasma proteins. This concentrate is then administered via injection.

ELIGIBILITY:
Inclusion Criteria:

* Female patient with mild to moderate SUI

Exclusion Criteria:

* Under anti-platelet agent treatment
* Platelet dysfunction syndrome
* Critical thrombocytopenia
* Acute and chronic infections
* Anti-coagulation therapy
* History of malignancy

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
urinary incontinence severity by PRP treatment | From baseline to 3 months after the PRP treatment day.
  Assessment of urinary incontinence severity by visual analog scale as: from 0 -10,

SECONDARY OUTCOMES:
Patients can control voiding on stress | From baseline to first month and continued to 3 months after the treatment day
  Assessment of the patient urine control status as daily pad use, maximum flow rate, and urine residual.

CONTACTS AND LOCATIONS:
Locations (1):
- SAYED GALAL HOSPITAL, AND AlGalaaTeaching HOSPITAL, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided